CLINICAL TRIAL: NCT07314047
Title: a Prospective, Multi-center, Open-label, Non-inferiority, Randomized, Controlled Registration Trial of the Liquid Embolic Agent for the Treatment of Brain Arteriovenous Malformation
Brief Title: The Liquid Embolic Agent for the Treatment of Brain Arteriovenous Malformation
Acronym: PARTNER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAVA-2023-01-CIP-00
Record Dates: First submitted 2025-01-16; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Brain Arteriovenous Malformation; Arteriovenous Fistula
Keywords: brain arteriovenous malformation; arteriovenous fistula; LIQUID EMBOLIC AGENT
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid embolic agent (Experimental): Liquid embolic agent developed and manufactured by MicroPort NeuroTech.Liquid embolic agents are used to embolize cerebrovascular malformations during the procedure.
  Interventions: Device: liquid embolic agent
- the Onyx Liquid Embolic System (Active Comparator): The Onyx Liquid Embolic System was developed and manufactured by Micro Therapeutics Inc. DBA ev3 Neurovascular. The Onyx Liquid Embolic System is used to embolize cerebrovascular malformations during the procedure.
  Interventions: Device: liquid embolic agent

INTERVENTIONS:
Device: liquid embolic agent — liquid embolic agent

SUMMARY:
This study is designed as a prospective, multi-center, open-label, non-inferiority, randomized controlled clinical trial. The control device is Onyx Liquid Embolic System marketed by Micro Therapeutics Inc. DBA ev3 Neurovascular (NMPA (J) 20173136690). According to the inclusion and exclusion criteria specified in this trial protocol, approximately 116 subjects with brain arteriovenous malformation will be enrolled for interventional embolization treatment. The subjects will undergo follow-up before the surgery, after device implantation, at discharge, 1 month (± 7 days), 6 months (± 30 days), and 12 months (± 60 days) after the first embolization. When necessary, unscheduled follow-up will be conducted to record various indicators for evaluating the safety and effectiveness of liquid embolic agents in the treatment of brain arteriovenous malformations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years at the time of signing the informed consent
* Subjects with brain arteriovenous malformation diagnosed by CT/MRI/DSA
* The target brain arteriovenous malformation is classified by Spetzler-Martin in the range of Ⅰ ~ Ⅳ
* Subjects themselves and/or their guardian are able to understand the purpose of the study, consent to participate, and sign the informed consent form
* Brain arteriovenous malformations deemed suitable for liquid embolic agent intervention as assessed by the investigator

Exclusion Criteria:

* Multiple brain arteriovenous malformations
* Brain arteriovenous malformation complicated with blood flow-related aneurysm that may require staged and delayed treatment using other methods within the one-year follow-up period
* Brain arteriovenous malformation with a history of stereotactic radiosurgery within 3 years
* Brain arteriovenous malformation with bleeding within 1 week
* Brain arteriovenous malformation with an expected number of embolizations ≥ 4
* Brain arteriovenous malformation scheduled for surgical resection after embolization
* mRS score ≥ 3
* Subjects unsuitable for anesthesia or endovascular surgical treatment, due to major diseases of cardio, lung, liver, spleen or kidney, malignant brain tumors, severe active infection, disseminated intravascular coagulation, or a history of severe mental illness, etc
* Subjects who undergo major surgical procedures (such as tumor resection, vital organ surgery, etc.) within 30 days prior to signing the informed consent form, or those scheduled for such procedures within 60 days after signing the informed consent form
* Contraindications for liquid embolic agent treatment, including but not limited to: contraindications for DSA, severe allergy or intolerance to contrast agents, severe allergy or intolerance to antiplatelet or anticoagulant medications required for treatment, or severe allergy to tantalum metal
* Pregnant or lactating women
* Subjects participating in other drug or device studies that have not reached their endpoints or who have just withdrawn from the group for less than one month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Rate of effective embolization of target brain arteriovenous malformation | Perioperative
  Effective embolization refers to a reduction of ≥ 50% after the last embolization of the target brain arteriovenous malformation compared with that before the first embolization

SECONDARY OUTCOMES:
Rate of favorable clinical outcomes during the 1 year follow-up period | 1 year after procedure
  Favorable clinical outcome refers to a mRS score of ≥ 0 and ≤ 2
Incidence of symptomatic stroke or death within one month after procedure | 1 month after procedure
Incidence of symptomatic intracranial hemorrhage related to procedure within 1 month after procedure | 1 month after procedure
Incidence of symptomatic ischemic stroke related to procedure within 1 month after procedure | 1 month after procedure
Incidence of device-related serious adverse events during the 1 year follow-up period | 1 year after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
To be decided